CLINICAL TRIAL: NCT00239187
Title: A Randomized, Double-blind, Placebo-controlled Clinical Trial to Evaluate the Safety, Tolerability, Pharmacokinetics and Clinical Response of Repeated Subcutaneous Doses of E1 in Combination With G1 in Patients With Type 2 Diabetes
Brief Title: A Study in Type 2 Diabetic Patients With Repeated Doses of E1 in Combination With G1
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: OPKO Health, Inc. (Industry)
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: INT-202
Record Dates: First submitted 2005-10-12; First posted 2005-10-14 (Estimated); Last update posted 2019-10-18 (Actual); Status verified 2019-10

CONDITIONS: Type 2 Diabetes
Keywords: Type 2 diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — methyl N-acetylsibirosaminide

INTERVENTIONS:
Drug: E1 and G1

SUMMARY:
The purpose of the study is to determine whether E1 and G1 are safe and effective in the treatment of type 2 diabetes.

Type 2 diabetes is the most common form of diabetes. The disease is characterised by insulin resistance and a compensated state of hyperinsulinemia. In most individual, hyperglycemia results from a failure of pancreatic beta cells insulin secretory capacity to adequately compensate for insulin resistance in peripheral tissues. Treatment for type 2 diabetes is achieved by dietary control, or a combination of diet and oral hypoglycemic agents or insulin. As the disease progress, many type 2 diabetic patients eventually require insulin as primary therapy to achieve glycemic control.

Recent diabetic research has increasingly focused on pancreatic islet cell replacement, either by islet cell transplantation or by endogenous regeneration of islet cells. During fetal development, islet precursor cells proliferate and differentiate into mature beta cells capable of producing insulin. This process is known as islet cell neogenesis. Islet cell neogenesis normally ceases around birth, however, the adult pancreas still retains significant potential for islet regeneration, as shown by tissue repair following pancreatic injury. Pre-clinical studies have shown that E1 and G1 can re-establish islet cell neogenesis and increase insulin production in diabetic animal models. In type 2 diabetic patients, treatment with E1 and G1 may result in islet cell regeneration. This therapeutic approach may improve beta cell function, restore the loss of insulin secretory capacity and also benefit patients on oral hypoglycemic agents by delaying insulin use.

DETAILED DESCRIPTION:
In this study, 30 type 2 diabetic patients requiring oral hypoglycemic therapy with Metformin and/or Thiazolidinedione will be randomized. Twenty (20) patients will be randomized to receive active study medication and 10 patients will be randomized to receive vehicle control. After undergoing screening procedures, potential patients will enter a 14 day baseline phase where baseline data will be collected. Pending successful completion of the baseline phase, patient will enter a 28-day treatment phase where they will be randomized to receive either once daily subcutaneous injections of E1 plus G1, as separate injections or once daily subcutaneous injections of vehicle control (as 2 separate injections). Patients will receive once daily doses in the morning after breakfast for a period of 28 days. Upon completion of treatment, all patients will continue in the follow-up phase for an additional 6 months and will return to the clinic for monthly visits. Throughout the study, patients will remain on their current oral hypoglycemic therapy with Metformin and/or Thiazolidinedione and will maintain a diary record of blood glucose levels.

The body's ability to control glucose will be assessed by oral glucose tolerance test (OGTT). After an overnight fast, patients will be asked to drink a solution containing a known amount of glucose. Blood samples for glucose and insulin measurements will be obtained before the patients drink the glucose solution, and again 30 minutes, 60 minutes and 2 hours after the glucose is consumed. This test will be performed at frequent intervals during the study.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent obtained from participants
* Clinical diagnosis Type 2 diabetes requiring treatment with Metformin and/or TZD and who are otherwise healthy
* On a stable Metformin and/or TZD regimen for at least 60 days prior to screening
* Maximum stimulated c-peptide level > 0.6 nmol/L (1.8 ng/mL)
* Currently self monitoring blood glucose levels (i.e. daily)
* No episodes of severe hypoglycemia for 60 days prior to screening
* Body mass index within the range 25-40 kg/m2
* Patient cannot live alone during the treatment phase and up to 1 month in follow-up

Exclusion Criteria:

* Known of suspected history of significant liver, or other GI disease
* History of significant cardiovascular disease including stroke, peripheral vascular disease or any related symptoms
* History of peptic ulcer disease and/or GI bleeding/perforation
* History of cancer
* History or presence of proliferative retinopathy, severe non-proliferative retinopathy, macular edema or presence of untreated diabetic eye disease
* History of treated peripheral or autonomic neuropathy
* Serum creatine superior or equal to 2.0 mg/dL
* Non-healed diabetic ulcer
* History of hypoglycemic unawareness

Ages: 30 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30
Dates: Start 2005-09; Study Completion 2007-01 (Actual)

PRIMARY OUTCOMES:
To assess the safety and tolerability of repeated subcutaneous doses of E1 in combination with G1 in patients with type 2 diabetes

SECONDARY OUTCOMES:
To evaluate the pharmacokinetics (PK) profile and clinical effects of repeated subcutaneous doses of E1 in combination with G1 in patients with type 2 diabetes

CONTACTS AND LOCATIONS:
Overall Officials: Aleksandra Pastrak, M.D., Study Director — OPKO Health, Inc.
Locations (3):
- United States (3):
  - Profil Institute for Clinical Research Inc., Chula Vista, California
  - Clinical Research of West Florida, Clearwater, Florida
  - Diabetes and Glandular Disease Research Associates, San Antonio, Texas